CLINICAL TRIAL: NCT02207192
Title: Effect of Weight Loss on Postural Changes in Pulmonary Function : a Longitudinal Study in Morbidly Obese to Obese Subjects Following Gastroplasty
Brief Title: Postural Changes in Lung Volumes in Obesity
Status: Completed | Type: Observational
Sponsor: Association pour la Formation du Personnel à la Medecine d'Urgence (Other)
Responsible Party: Sponsor
Other Study IDs: FRC obesity
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Obesity
Keywords: obesity, lung volumes, postural changes
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Morbidly obese: Consecutive morbidly obese adults (BMI over or equal to 40 kg/m2) scheduled for bariatric surgery were prospectively recruited.Subjects with respiratory and cardiac history (asthma, Chronic obstructive pulmonary disease, heart failure) were excluded.
  Interventions: Other: Postural change in lung volumes: sitting to Supine

INTERVENTIONS:
Other: Postural change in lung volumes: sitting to Supine — Pulmonary function and arterial blood gases were assessed both prior to and after weight loss as part of pre-operative and 12-month follow-up evaluations.
  Pulmonary function tests were performed both in the sitting and then in the supine position.

SUMMARY:
Postural changes are known to affect normal lung volumes. A reduction in sitting to supine functional residual capacity (FRC) is well-described in non-obese subjects adopting a supine position. However, postural changes in lung volumes in the obese require further exploration. We aimed to longitudinally address the effects of weight loss on postural changes in lung volumes and pulmonary function, in obesity. We tested the hypothesis that supine reduction in FRC would be absent in morbid obesity and recovered upon weight loss.

ELIGIBILITY:
Inclusion Criteria:

* subjects scheduled for bariatric surgery (BMI over or equal to 40 kg/m2)

Exclusion Criteria:

* Subjects with respiratory and cardiac history (asthma, COPD, heart failure) were excluded.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Twelve morbidly obese adults (BMI over or equal to 40 kg/m2) scheduled for bariatric surgery at the Montpellier university hospital were recruited. They were 3 men and 9 women.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2005-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
functional residual capacity | baseline and one year after bariatric surgery

SECONDARY OUTCOMES:
lung volumes and flows | at baseline and after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Sebbane, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University hospital, Montpellier, France

REFERENCES:
- [Derived] Sebbane M, El Kamel M, Millot A, Jung B, Lefebvre S, Rubenovitch J, Mercier G, Eledjam JJ, Jaber S, Hayot M. Effect of Weight Loss on Postural Changes in Pulmonary Function in Obese Subjects: A Longitudinal Study. Respir Care. 2015 Jul;60(7):992-9. doi: 10.4187/respcare.03668. Epub 2015 Apr 7. PMID 25852166